CLINICAL TRIAL: NCT02860546
Title: A Phase 2 Study With Safety Lead-in, Evaluating TAS-102 Plus Nivolumab in Patients With Microsatellite Stable Refractory Metastatic Colorectal Cancer
Brief Title: A Study Evaluating TAS-102 Plus Nivolumab in Patients With MSS CRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS-102-203
Record Dates: First submitted 2016-07-13; First posted 2016-08-09 (Estimated); Results first posted 2021-07-26 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Refractory Metastatic Colorectal Cancer
Keywords: Refractory; Metastatic; Colorectal cancer; TAS-102; Nivolumab; Microsatellite Stable; Programmed cell death protein1 (PD 1)
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — trifluridine tipiracil drug combination; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS-102 + Nivolumab (Experimental): Participants received a dose of 35 milligrams per meter square (mg/m^2) of TAS-102 tablets orally twice per day (BID) within 1 hour after completion of morning and evening meals, in 4-week cycle. In each 4-week cycle, TAS-102 was administered for 2 weeks, as 5 days a week with 2 days rest, followed by a 14-day rest. Also participants received 3 milligrams per kilogram per dose (mg/kg/dose) Nivolumab intravenous (I.V) infusion over 60 minutes every 14 days (on Day 1 and Day 15 of each 4-week cycle).
  Interventions: Drug: TAS-102; Drug: nivolumab

INTERVENTIONS:
Drug: TAS-102 — One Arm Only (of TAS 102 plus nivolumab)
  Other Names: Lonsurf®
Drug: nivolumab — One Arm Only (of TAS 102 plus nivolumab)
  Other Names: Opdivo®

SUMMARY:
A Phase 2 Study with Safety Lead-in, Evaluating TAS-102 Plus Nivolumab in Participants with Microsatellite Stable Refractory Metastatic Colorectal Cancer

DETAILED DESCRIPTION:
This is a multicenter, single arm, safety lead-in, Phase 2 study, using Simon's 2 stage design evaluating the safety and efficacy of TAS-102 plus nivolumab in participants with Microsatellite-stable refractory metastatic colorectal cancer

Stage 1: Participants will be enrolled and after Cycle 1 treatment, they will be evaluated for the safety and tolerability of the combination therapy. Assuming a tolerated dose is confirmed additional participants evaluable for response will be enrolled and followed for a minimum of 6 months and there will be an interim analysis to assess the safety and efficacy to determine whether the second stage will open for enrollment.

Stage 2: Additional participant evaluable for response assessment will be enrolled and followed for a minimum of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent.
2. Participants with confirmed histologically proven metastatic or locally advanced colorectal adenocarcinoma who are microsatellite stable (MSS) (ie, not microsatellite instable [MSI]) based on either an analysis of tissue from a prior biopsy or based on tissue from a new biopsy.
3. Participants with the presence of at least 1 lesion with measurable disease as defined by 10 millimeters (mm) in the longest diameter for a soft tissue lesions or 15 mm in the short axis for a lymph node by response evaluation criteria in solid tumors (RECIST) and immune related response-criteria (irRC) for a response assessment.
4. Participants has received at least 2 prior lines of standard chemotherapies for metastatic colorectal cancer (mCRC) and is refractory to or failing those chemotherapies.
5. Age greater than or equal to (>=) 18 years.
6. Eastern Cooperative Oncology Group performance status of 0 to 1
7. Life expectancy of >=4 months.
8. Has adequate organ function.
9. Women of childbearing potential must have a negative pregnancy test (urine or serum) within 7 days before starting study drugs. Is able to take medications orally.
10. Is able to take medications "orally".

Exclusion Criteria:

1. Has a serious illness or medical condition.
2. Treatment with any of the following within the specified time frame before enrollment:

   1. Major surgery within the past 4 weeks (the surgical incision should be fully healed before study drug administration).
   2. Any anticancer therapy within the past 3 weeks before enrollment.
   3. Extended field radiation within the past 4 weeks or limited field radiation within the past 2 weeks before enrollment.
   4. Any investigational drug/device received within the past 4 weeks or 5 times the half-life (whichever is shorter) before enrollment.
3. Previous treatment with TAS-102.
4. Prior treatment with anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death ligand (anti-PD-L1), anti programmed cell death ligand 2, anti-CD137, anti-OX-40, anti CD40, anti cytotoxic T lymphocyte associated antigen-4 antibodies, or any other immune checkpoint inhibitors.
5. Unresolved toxicity of >=Common Terminology Criteria for Adverse Events version (CTCAE) version 4.03 grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum induced neurotoxicity).
6. Prior events of immune-mediated pneumonitis, immune-mediated colitis, immune-mediated hepatitis, immune-mediated endocrinopathies, immune mediated nephritis and renal dysfunction, immune mediated rash, immune mediated encephalitis, and history of infusion reactions to nivolumab.
7. Known or assumed hypersensitivity to TAS-102 or nivolumab or any of its ingredients, including polysorbate 80-containing infusion.
8. Previous severe hypersensitivity reaction to treatment with another mAb.
9. Pregnant or lactating female.
10. Inappropriate for entry into this study in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Study results using compiled efficacy and safety data will be published at congress or to a journal, without any identification of the patients.

REFERENCES:
- [Derived] Patel MR, Falchook GS, Hamada K, Makris L, Bendell JC. A phase 2 trial of trifluridine/tipiracil plus nivolumab in patients with heavily pretreated microsatellite-stable metastatic colorectal cancer. Cancer Med. 2021 Feb;10(4):1183-1190. doi: 10.1002/cam4.3630. Epub 2021 Feb 5. PMID 33544407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centers in United States.
Pre-assignment Details: A total of 22 participants were screened out of which 18 participants passed the screening and were enrolled in the study. This study was planned to have 2 stages but only stage1 was completed. The study was halted following an interim analysis and no participants were enrolled in stage 2. Therefore, the data represented is for stage 1 only.
Period: Overall Study
Arm/Group | TAS-102 + Nivolumab
Started | 18
Completed | 0
Not Completed | 18
Not completed — Clinical Progression | 6
Not completed — Radiological Progression | 12

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- TAS-102 + Nivolumab: Participants received a dose of 35 mg/m^2 of TAS-102 tablets orally BID within 1 hour after completion of morning and evening meals, in 4-week cycle. In each 4-week cycle, TAS-102 was administered for 2 weeks, as 5 days a week with 2 days rest, followed by a 14-day rest. Also participants received 3 mg/kg/dose Nivolumab I.V infusion over 60 minutes every 14 days (on Day 1 and Day 15 of each 4-week cycle).
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Immune-Related Overall Response Rate (irORR)
Description: irORR was defined as the percentage of participants achieving a complete response (irCR) or partial response (irPR) based on irRC criteria. Per irRC criteria, Complete Response (irCR) was defined as the disappearance of all tumor lesions (measurable or not, and no new lesions)., Partial Response (irPR) was defined as a decrease in the sum of the products of the two largest perpendicular diameters (SPD) by 50 percent (%) or greater by a consecutive assessment at least 4 weeks after first documentation, Stable Disease (irSD) was defined as the failure to meet criteria for irCR or irPR in absence of progressive disease (irPD), irPD was defined as at least 25% increase in SPD relative to nadir.
Time Frame: From first dose of study treatment up to 30 days after the last dose of study treatment (up to 53 weeks)
Population: Efficacy population included all participants in the safety population (all participants who received at least 1 dose of study drug) who completed at least 6 months of tumor follow-up, unless the participant progressed or died before the 6-month follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
percentage of participants | 0

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT: defined as occurrence of any of the following-
  Hematological toxicities:
  * Grade 4 neutropenia lasting greater than(>)7 days
  * Grade 4 febrile neutropenia and fever greater than or equal to (>=)38 degree celsius for over 1 hour
  * Grade 4 thrombocytopenia or grade 3 thrombocytopenia associated with bleeding or requiring transfusions
  Non-hematological toxicities:
  * Grade 3 or grade 4 non-hematologic toxicity (excluding alopecia, nausea, vomiting, diarrhea)
  * Grade 3 or grade 4 nausea/vomiting lasting >48 hours and uncontrolled by aggressive anti-emetic therapy, including serotonin 5-HT3 receptor antagonists (e.g, ondansetron)
  * Grade 3 or grade 4 diarrhea lasting > 48 hours and unresponsive to antidiarrheal medication
  Drug-related toxicities:
  * Any drug-related toxicity resulting in > 2 weeks delay in initiation of Cycle 2 (i.e, cannot start Cycle 2 until Day 43 or later)
  * Any drug-related toxicity that prevents completion of 80% compliance for either drug in Cycle 1
Time Frame: Cycle 1 (each cycle is of 4 weeks)
Population: DLT Evaluable (DLTE) population included all participants in the safety population in Stage 1, prior to confirming the recommended dose, who completed at least 1 cycle (28 days) of study treatment with at least 80% of the study treatment administered, unless the treatment was interrupted because of a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Recommended Phase 2 Dose (RP2D)
Description: RP2D of TAS-102 was evaluated based on the safety and tolerability of the combination therapy of TAS-102 and Nivolumab.
Time Frame: Cycle 1 (each cycle is of 4 weeks)
Population: DLTE population included all participants in the safety population in Stage 1, prior to confirming the recommended dose, who completed at least 1 cycle (4 weeks) of study treatment with at least 80% of the study treatment administered, unless the treatment was interrupted because of a DLT.
Measure: Number; unit: mg/m^2
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 6
mg/m^2 | 35

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical condition that occurs in a participants while participating in a clinical study and does not necessarily have a causal relationship with the use of the study treatment. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs: AEs that developed or worsened during the on-treatment period which was defined as the period from the time of first dose of study treatment until 30 days after the last dose of study treatment.
Time Frame: From first dose of study treatment up to 30 days after the last dose of study treatment (up to 53 weeks)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
participants
  Participants with TEAEs | 18
  Participants with TESAEs | 6

5. Secondary Outcome: Number of Participants With Grade 3 or Higher Laboratory Tests Abnormalities
Description: Hematological and chemistry laboratory tests abnormalities were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. as: Grade 1 (Mild, asymptomatic or mild symptoms); Grade 2 (Moderate, minimal, local or noninvasive intervention indicated); Grade 3 (Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated); Grade 4 (Life-threatening consequences, urgent intervention indicated); Grade 5 (Death related to AE).
Time Frame: From first dose of study treatment up to 30 days after the last dose of study treatment (up to 53 weeks)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
participants
  Grade 4: Neutropenia (neutrophils low) | 3
  Grade 4: Anemia (hemoglobin low) | 1
  Grade 4: Leukopenia (leukocytes low) | 0
  Grade 4: Lymphopenia (lymphocytes low) | 0
  Grade 4: Thrombocytopenia (platelets low) | 0
  Grade 4: Bilirubin High | 0
  Grade 4: Glucose High | 0
  Grade 4: Sodium Low | 0
  Grade 3: Neutropenia (neutrophils low) | 3
  Grade 3: Anemia (hemoglobin low) | 1
  Grade 3: Leukopenia (leukocytes low) | 6
  Grade 3: Lymphopenia (lymphocytes low) | 2
  Grade 3: Thrombocytopenia (platelets low) | 1
  Grade 3: Bilirubin High | 1
  Grade 3: Glucose High | 1
  Grade 3: Sodium Low | 1

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with objective evidence of complete response (CR) or partial response (PR) per response evaluation criteria in solid tumors (RECIST) version 1.1.CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than (<)10 millimeters (mm). PR was defined as at least a 30 % decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters.
Time Frame: From first dose of study treatment up to 30 days after the last dose of study treatment (up to 53 weeks)
Population: Efficacy population included all participants in the safety population who completed at least 6 months of tumor follow-up, unless the participant progressed or died before the 6-month follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
percentage of participants | 0

7. Secondary Outcome: Progression-Free Survival (PFS) Based on Immune Related Response-Criteria (irRC)
Description: Immune-related progression free survival was defined as the time (in months) from the date of first dose of study treatment until the date of the investigator-assessed radiological disease progression (based on irRC) or death due to any cause. Participants who were alive with no disease progression at the moment of the analysis cut-off date was censored at the date of the last tumor assessment. Per irRC criteria disease progression defined as at least 25% increase in SPD relative to nadir. Analysis was performed using Kaplan-Meier estimates.
Time Frame: From the first dose of study treatment to disease progression or death (up to 53 weeks)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
months
  Radiologic progression of disease only | 2.2 [1.8 to 6.0]
  Radiologic + clinical progression of disease | 2.2 [1.8 to 3.7]

8. Secondary Outcome: Progression-Free Survival (PFS) Based on RECIST Criteria
Description: Progression free survival was defined as the time (in months) from the date of first dose of study treatment until the date of the investigator-assessed radiological disease progression (based on RECIST 1.1) or death due to any cause. Per RECIST criteria disease progression defined as least 20% increase in the sum of diameters of the target lesions, taking as a reference the smallest sum on study, including the baseline sum. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Definitive new lesion presence also indicated progression.
Time Frame: From the first dose of study treatment to disease progression or death (up to 53 weeks)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
months
  Radiologic progression of disease only | 2.8 [1.8 to 5.1]
  Radiologic + clinical progression of disease | 2.5 [1.8 to 3.7]

9. Secondary Outcome: Disease Control Rate (DCR) Based on irRC Criteria
Description: DCR was defined as the percentage of participants with objective evidence of radiologic complete response (CR), partial response (PR), or stable disease (SD) and was based on the overall best response from each participant as determined from investigator response assessments and following irRC criteria. Per irRC criteria, CR was defined as the disappearance of all tumor lesions (measurable or not, and no new lesions). PR was defined as a decrease in the sum of the products of the two largest perpendicular diameters by 50% or greater by a consecutive assessment at least 4 weeks after first documentation. SD was defined as the failure to meet criteria for irCR or irPR in absence of in absence of irPD.
Time Frame: From first dose of study treatment up to 30 days after the last dose of study treatment (up to 53 weeks)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
percentage of participants | 44.4 [21.5 to 69.2]

10. Secondary Outcome: Disease Control Rate (DCR) Based on RECIST Criteria
Description: DCR was defined as the percentage of participants with objective evidence of radiologic CR, PR, or SD and was based on the overall best response from each participant as determined from investigator response assessments and following RECIST Criteria version 1.1. Per RECIST Criteria CR defined as disappearance of all target lesions. Reduction in any pathological lymph nodes in short axis to <10 mm. PR defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as a reference the smallest sum diameters during study.
Time Frame: From first dose of study treatment up to 30 days after the last dose of study treatment (up to 53 weeks)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 18
percentage of participants | 55.6 [30.8 to 78.5]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of the study treatment to the death in the safety population. Participants alive at the time of the study discontinuation were censored. Analysis was performed using Kaplan-Meier estimates.
Time Frame: From first dose of study treatment up to 30 days after the last dose of study treatment (up to 53 weeks)
Population: Safety population included all participants who received at least 1 dose of study drug. Overall number of participants analyzed is 0 because data were not collected for the outcome measure at particular time point.
Arm/Group | TAS-102 + Nivolumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 30 days after the last dose of study treatment (up to 53 weeks)
Description: Analysis was performed on safety population.
Arm/Group | TAS-102 + Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 6/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102 + Nivolumab (N=18)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (3)
Pyrexia (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102 + Nivolumab (N=18)
Anaemia (Blood and lymphatic system disorders) | 5 (11)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Photopsia (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 11 (22)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (25)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (9)
Asthenia (General disorders) | 2 (2)
Fatigue (General disorders) | 6 (14)
Mucosal inflammation (General disorders) | 2 (6)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Candida infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Medication error (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 6 (14)
Platelet count decreased (Investigations) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash follicular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
After interim analysis, per study design plan, the trial was stopped for futility before enrollment into Stage 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT02860546/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/46/NCT02860546/SAP_001.pdf